CLINICAL TRIAL: NCT04230967
Title: Ambulation for Latency During Expectant Management of PPROM: A Randomized Controlled Trial (AMBLE)
Brief Title: Ambulation for Latency During Expectant Management of PPROM
Acronym: AMBLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Fitbit Health Solutions (Unknown); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Beth Leong Pineles, Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-19-0982
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Preterm Premature Rupture of the Membranes; Pregnancy Complications; Pregnancy, High Risk
Keywords: pregnancy; PPROM
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Pregnancy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambulation Group (Experimental): Participants in the ambulation arm will be allowed ad lib activity and instructed that they should walk at least once per day out of their room with a goal of 2,000 steps per day. The Fitbit InspireTM devices will be set to this goal and notifications will be given on the device for the participants meeting their goals. Upon enrollment, they will be given a pamphlet with instructions to ambulate out of the room at least once per day with a goal of 2,000 steps daily and their Fitbits will be pre-programmed with this goal. Study staff will also remind participants to ambulate via email, text or in-person if they are not meeting their goal of 2,000 steps per day.
  Interventions: Behavioral: Ambulation Group
- Routine Care (Active Comparator): Participants in the routine care arm will be allowed ad lib activity but no encouragement to walk will be given. They will not have any goals set on their Fitbits. Upon enrollment, they will be given pamphlets with no instruction on whether or not to ambulate and their Fitbits will be pre-programmed to have no goal.
  Interventions: Behavioral: Routine Care

INTERVENTIONS:
Behavioral: Ambulation Group — Participants in the ambulation arm will be allowed ad lib activity and instructed that they should walk at least once per day out of their room with a goal of 2,000 steps per day. The Fitbit Inspire devices will be set to this goal and notifications will be given on the device for the participants meeting their goals
  Arms: Ambulation Group
Behavioral: Routine Care — No encouragement to ambulate will be provided to subjects. Their movement will be recorded
  Arms: Routine Care

SUMMARY:
Ambulation in pregnancy has been proposed to decrease stress and anxiety, increasing preterm birth. Whether ambulation is causally related to latency is unknown. The FitBit will be used for tracking the number of steps taken daily by each participant, and for encouraging the intervention group to walk. The FitBit is the most widely used physical activity tracker in medical research, and its use has been validated for research use in pregnant women. The purpose of the study is to evaluate whether ambulation in patients with preterm premature rupture of the membranes (PPROM) prolongs latency.

ELIGIBILITY:
Inclusion Criteria

* Pregnant women aged 12-55
* Gestational age 23 0/7 to 35 0/7 weeks
* PPROM confirmed by clinical diagnosis which includes sterile speculum examination with pooling, ferning, and nitrazine tests, or the Amnisure ROM Test
* Planned inpatient expectant management with delivery goal >=7 days from enrollment
* Ability to provide informed consent in English or Spanish

Exclusion Criteria

* Imminent delivery
* Transverse or footling breech presentation (if multiple gestation, presenting fetus)
* Unstable lie (if multiple gestation, presenting fetus)
* Funic presentation (if multiple gestation, presenting fetus)
* Active vaginal bleeding
* Regular, painful contractions (>=3 in 10 minutes for 30 minutes or more) consistent with labor
* Clinical contraindication to ambulation as determined by the managing physician
* Physician declines to have the patient approached for participation
* Lethal fetal anomalies

Ages: 12 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Latency (measured in days) from from randomization to delivery | 12 weeks

SECONDARY OUTCOMES:
Maternal Infectious morbidity | at delivery
  Chorioamnionitis, endometritis
# of subjects with Placental abruption | at delivery
# of subjects with Cesarean delivery (and emergent cesarean delivery) | at delivery
# of subjects with Umbilical cord prolapse | at delivery
# of subjects with Maternal venous thromboembolism | at delivery
Maternal Readmission | within 6 weeks of delivery- 6 weeks
Time to delivery (time-to-event outcome) | 12 weeks
Delivered at >7 days post randomization | at delivery
Maternal antepartum hospitalization length of stay | from admission to delivery
Measurement of Stress outcomes utilizing Perceived Stress Scale (PSS) | 7 days
  comparison between 2 groups- as measured by validated Stress survey. Scaled 0-4 corresponding response of Never to very often respectively. Change from baseline to day 7
Measurement of Anxiety outcomes utilizing State Trait Anxiety Inventory (STAI) | 7 days
  comparison between 2 groups-as measured by validated anxiety survey. Scaled 1-4 corresponding response of Not at all to very much so. Change from baseline to day 7
Measurement of Depression outcomes utilizing Edinburgh Depression Scale (EDS) | 7 days
  comparison between 2 groups-as measured by validated depression scale. Maximum score: 30 Possible Depression: 10 or greater Always look at item 10 (suicidal thoughts) Change from baseline to day 7
Measurement of Patient Satisfaction by validated satisfaction survey between 2 groups | at delivery
  comparison between 2 groups-as measured by validated survey from the last questionnaire answered prior to delivery
Fetal or neonatal death | at discharge
Apgar score < 5 at 5 minutes of life | at delivery
Umbilical arterial pH < 7.00 | at delivery
# of neonates with Small for gestational age | at delivery
  defined as < 5th percentile weight for gestational age, assessed specifically by sex and race of the infant based on United States birth certificate data
# of neonates with Neonatal intraventricular hemorrhage (IVH) grades III or IV | at discharge
  as determined by cranial ultrasounds performed as part of routine clinical care and classified based on the Papule classification system
# of neonates with Neonatal periventricular leukomalacia (PVL) | at discharge
# of neonates with Neonatal necrotizing enterocolitis (NEC) | at discharge
# of neonates with Neonatal retinopathy of prematurity (ROP). | at discharge
  This diagnosis will be reached when an ophthalmologic examination of the retina has been performed and ROP is diagnosed at Stage I (demarcation line in the retina) or greater.
# of neonates with Bronchopulmonary dysplasia (BPD) | at discharge
  defined as oxygen requirement at 28 days of life or at 36 weeks postmenstrual age for infants born before 32 weeks.
Gestational age at delivery < 28 weeks | at delivery
Gestational age at delivery < 34 weeks | at delivery
Neonatal length of hospital stay, based on admission to NICU or intermediate care unit | at discharge
Composite adverse maternal outcome (CMAO) | at discharge
Composite adverse fetal/neonatal outcome | at discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Universtiy of Texas Health Science Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No